CLINICAL TRIAL: NCT05164874
Title: Evaluation of a Mobile Mammography Unit. A Randomized Cluster Trial Protocol of a Population Health Intervention Research to Reduce Breast Cancer Screening Disparities in Normandy, France (Mammobile)
Brief Title: A Randomized Cluster Trial to Evaluate a Mobile Mammography Unit in Breast Cancer Screening in France (Mammobile)
Acronym: Mammobile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Université de Caen Normandie (Other)
Collaborators: National Cancer Institute, France (Other Government); Regional health agency, Normandy France (Unknown); Pink ribbon (Ruban Rose, France) (Unknown); Normandy regional cancer screening coordination center (Unknown); Departmental councils (Unknown)
Responsible Party: Principal Investigator, Élodie Guillaume, PhD in Epidemiology and Public Health, Université de Caen Normandie
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UCaenNormandie
Record Dates: First submitted 2021-12-03; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: breast cancer screening; mobile mammography unit; social and territorial inequalities; randomized cluster trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This intervention will be conducted as a prospective randomized controlled cluster trial.The cluster of the study is an aggregation of géographical areas. It was done according to the travel time to the radiology centres, the most distant areas has been selected and then merged with neighbouring areas, still by distance run, until reaching areas of the expected population size. This except size is around 100 women. Expecting a 40% participation to the mobile unit, we will achieve 32 to 48 mammograms daily. A randomization in parallel group have been perform to constitute the intervention arm and the control arm.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Women will receive a proposition for an appointment at the MMU in complement to the current screening invitation, keeping the choice of their place of screening.
  Women will also receive the timetable of prevention actions with the invitation to participate in screening.
  Interventions: Device: Mobile Mammography Unit
- Control (No Intervention): No change from the usual breast cancer screening organization

INTERVENTIONS:
Device: Mobile Mammography Unit — The main intervention will be a proposition for an appointment at the MMU in complement to the current OBCS
  Arms: Intervention

SUMMARY:
Organized breast cancer screening (OBCS) has been implemented nationwide since 2004 inFrance, but the participation rate remains low (51%) and inequities in participation were reported. Strategies as mobile mammography units could be effective to increase participation in OBCS and reduce inequities, especially in underserved areas in regard to this screening. Our main objective is to evaluate this device and to identify how to incorporate a mobile unit in the OBCS with a view to tackle territorial inequities in OBCS participation. The project will be conducted as a randomized controlled cluster trial in 2022-2024, in remote areas of 4 French departments. The main intervention is to propose an appointment at the mobile unit in complement to the current OBCS in these remote areas. In addition, few weeks before this intervention, local actors will carry out actions to promote OBCS with mobile unit specific information tools. This randomized controlled trial will provide a high level of evidence in assessing the mobile unit effects on participation and inequities.

DETAILED DESCRIPTION:
Context In most EU member states, breast cancer screening is organised with a mammography screening. However, there are still differences in the way screening programmes are implemented. In France, the organized breast cancer screening (OBCS) has been conducted, nationwide since 2004. A screening mammography is offered every two years to women aged 50 to 74 at average risk for this cancer. They receive from management structures in charge of this screening (SMS), an invitation to visit an accredited radiologist's office. A radiological imaging of the breast with two views plus a clinical breast examination is realized. Two different radiologists assure readings. In the last three year, the national participation rate remains stable around 51%. In addition, studies, using ecological indices of deprivation, highlight social and territorial inequalities: women living in disadvantaged area or far from a radiologist's office less participate. Different strategies can be implemented to increase participation to breast cancer screening, especially in populations with low-income or in rural areas, who have less access to screening. Among these strategies, mobile mammography units (MMU) seem effective. Therefore, in the French context, there is very little evidence on how to intervene to reduce health socio-territorial inequalities in screening, so public health decision-makers are unable to base proposals on evidence.

Intervention The main intervention will be a proposition for an appointment at the MMU in complement to the current OBCS. This complementary mode of screening offers the possibility for women furthest away from the radiologist's office to undergo screening in the MMU. All women eligible for OBCS and living in the zone selected for the intervention will be invited to participate either in a radiologist's office or in the MMU, keeping the choice of their place of screening. The breast screening in the MMU will follow the same protocol as screening at the radiologist's office according to national recommendations, so that the quality level of screening proposed in the MMU will the same as in any radiologist office. The MMU will be equipped with a latest-generation digital scenographer as well as an ultrasound system according to the compliance rules of the specifications published by the National Institute of Cancer. The quality of the mammographic radiographic equipment will also be certified by the Nuclear Safety Agency.

About two weeks before the MMU is parked, local actors, will carry out actions to inform women on the organized breast cancer screening and on the MMU. Women will receive the timetable of these actions with the invitation to participate in screening.

Design This intervention will be conducted during two years in 2022-2024, as a prospective randomized controlled cluster trial in the general population in the departments of Calvados, Manche, Eure and Seine-Maritime (Normandy Region in the north west of France). The cluster of the study is a group of IRIS (Ilots Regroupés pour l'Information Statistique). This geographical unit is the smallest scale for which census data are available and represents an average of 2000 inhabitants.

An algorithm was developed to constitute clusters integrating some constraints in a regional scenario.

Aggregation of IRIS was done according to the travel time to the radiology centres, the most distant IRIS has been selected and then merged with neighbouring IRIS, still by distance run, until reaching areas of the expected population size. This except size is around 100 women. Expecting a 40% participation to the MMU, 32 to 48 mammograms daily should be performed.

This algorithm was applied to all IRIS according to distance rank, until no more aggregation was possible. 91,982 women (95.6%) and 1,067 IRIS (94.3%) were selected in the final population in 356 clusters (with 258 created by the algorithm).

All the women constituting the target population is geolocated and geocoded. Thus, for each woman, history of screening, the current date of screening invitation, IRIS of residence, level of social deprivation according to an ecological deprivation index (the European Deprivation Index) and the distance between the woman's house and the nearest approved radiologist's office are known.

A randomization in parallel group have been perform to constitute the intervention arm (n=178 clusters) and the control arm (n=178 clusters), corresponding to 45275 in intervention arm vs 46707 in control arm.

Evaluations The overall objectives of the study are to evaluate the intervention's ability a) to reduce the socio-territorial inequalities of participation in breast cancer screening in a regional area (Normandy) in setting remote from radiologist's office b) to increase participation rate and c) understand how intervention interact with contextual factors and which causal mechanisms leading to these results in order to identify the optimal modalities for extending the MMU at the national level.

Concerning the first two objectives, the main evaluation criterion will be participation in screening, measured and compared between the "intervention" and "control" arm, at the aggregate level (cluster) and individual level in intent to treat. At the aggregate level, the comparison of screening participation will allow us to measure the raw and age-standardized increase in participation due to the intervention. At the individual level, multilevel logistic regressions, taking into account cluster data, allow to assess the increase in the probability of participating in screening after adjustment of the social deprivation, age and other available individual characteristics.

Although the calculation of the number of subjects in the study came from a pragmatic approach, the intraclass correlation factor was estimated at 0.0083, which with an average area size of 318.6 women gives a design effect equal to 3.63. Thus, the minimum significant difference in participation that can be proven will be 1.5%.

Actors information action, will be prospectively registered in a dedicated database and will be include in the global model analysis.

To furthermore explore contextual effect and to provide elements of knowledge on the causal mechanisms contributing to the effectiveness of the intervention the quantitative analyses will be completed by a qualitative approach inspired by the combined approaches that have emerged in realistic randomised controlled trials, using a theory that goes beyond logic models to describe contextual mechanisms and contingencies. An intervention theory was developed and three auto questionnaires will respectively explore, the informed choice, satisfaction to realized the mammography in the mammobile and the ComB Model construct implied in the screening behaviour.

ELIGIBILITY:
Inclusion Criteria:

* women eligible to breast cancer screening campaign : aged 50 to 74 years, and with the only risk of breast cancer being age. The previous screening mammography dating from 22 months

Exclusion Criteria:

* outside the ages
* with specific risk of breast cancer

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91982 (Estimated)
Dates: Start 2022-02-14 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Aggregated breast cancer screening participation rate 3 months after the last invitation | 3 months after the last invitation at the end of the two years of the intervention
  Participation rate will be measure at area level and compare between intervention and control arm.
Individual breast cancer screening participation rate 3 months after the last invitation | 3 months after the last invitation at the end of the two years of the intervention
  It will also be assessed at indivdual level with multilevel logistic regression
Impact of the mobile unit on social inequalities in screening participation | 3 months after the last invitation at the end of the two years of the intervention
  Impact of the mobile mammography unit on social inequalities will be assessed by comparing intervention and control arm. Social statut is measure with an ecological deprivation index
Impact of the mobile unit on territorial inequalities in screening participation | 3 months after the last invitation at the end of the two years of the intervention
  impact of the mobile mammography unit territorial inequalities will be assessed by comparing intervention and control arm. The distance to the radiologiste center will be used as territorial mesure

SECONDARY OUTCOMES:
Informed choice to breast cancer screening for participating women | through study completion, an average of 3 month
  An autoquestionnaire adressed to control and intervention arm will compare the informed choice
Informed choice to breast cancer screening for non-participating women | Women will be considered as "non participating" 18 month after the invitation
  An autoquestionnaire adressed to control and intervention arm will compare the informed choice
Satisfaction to mammography | through study completion, an average of 3 month
  An autoquestionnaire adressed to control and intervention arm will adressed the satisfaction to the mammography screening
Com-B Model Evaluation for participating women | through study completion, an average of 3 month
  An autoquestionnaire adressed to control and intervention arm will assessed if the mobile mammography unit and the prevention action have been facilitators to opportunity, motivation or capacity, to participate to breast cancer screening
Com-B Model Evaluation for non-participating women | Women will be considered as "non participating" 18 month after the invitation
  An autoquestionnaire adressed to control and intervention arm will assessed if the mobile mammography unit and the prevention action have been facilitators to opportunity, motivation or capacity, to participate to breast cancer screening

CONTACTS AND LOCATIONS:
Overall Officials: Elodie Guillaume, PhD, Principal Investigator — Université de Caen Normandie
Locations (1):
- Normandy, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Yes
Individual data is collected as part of the usual organization of organized breast cancer screening. It is the authorized structure that manages these data.
Time Frame: Data concerning participation, place of participation, date, distance and socioeconomic status will be anonimously analysed after the two years.

REFERENCES:
- [Derived] Guillaume E, Rollet Q, Launay L, Beuriot S, Dejardin O, Notari A, Crevel E, Benhammouda A, Verzaux L, Quertier MC, Launoy G. Evaluation of a mobile mammography unit: concepts and randomized cluster trial protocol of a population health intervention research to reduce breast cancer screening inequalities. Trials. 2022 Jul 8;23(1):562. doi: 10.1186/s13063-022-06480-w. PMID 35804417